CLINICAL TRIAL: NCT02284230
Title: Glycaemic and Cardiovascular Efficacy of Liraglutide in Prediabetic Patients With End-stage Renal Disease
Brief Title: The Effect of Liraglutide in Patients With Prediabetes and Kidney Failure
Acronym: LiRA2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to recruit participants
Sponsor: Bo Feldt-Rasmussen (Other)
Collaborators: Novo Nordisk A/S (Industry); The GCP unit at Copenhagen University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Bo Feldt-Rasmussen, Professor, MD, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1149-7801
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Failure, Chronic; Prediabetic State
MeSH Terms: conditions — Kidney Failure, Chronic; Prediabetic State | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide treatment (Active Comparator): Subcutaneous, once daily injection of liraglutide, individually dosed up to 1.8 mg/day.
  Interventions: Drug: Liraglutide
- Placebo treatment (Placebo Comparator): Subcutaneous, once daily injection of placebo, individually dosed up to 1.8 mg/day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide
  Other Names: Victoza
  Arms: Liraglutide treatment
Drug: Placebo
  Arms: Placebo treatment

SUMMARY:
The present study will examine the effects of liraglutide treatment during 26 weeks on several cardiovascular risk factors in patients with prediabetes and end-stage renal disease (ESRD). The primary objective is to determine the efficacy of the treatment on glucose tolerance evaluated during a 3h 75g-oral glucose tolerance test (OGTT). Secondary objectives include various clinical and biochemical cardiovascular and safety parameters.

We hypothesise that treatment with liraglutide can improve glucose tolerance in prediabetic patients with ESRD by normalizing plasma glucose excursions during an OGTT and ameliorate other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease treated with chronic maintenance dialysis (haemodialysis or peritoneal dialysis)
* Impaired glucose tolerance (2h plasma glucose ≥ 7,8 and < 11.1 mmol/l following a 75g-OGTT) and/or impaired fasting glucose (fasting plasma glucose ≥ 6.1 and < 7.0 mmol/l) evaluated at the screening visit

Exclusion Criteria:

* Diabetes mellitus type 1 or type 2 (diagnose according to WHO criteria)
* Chronic pancreatitis / previous acute pancreatitis
* Known or suspected hypersensitivity to trial product(s) or related products
* Treatment with oral glucocorticoids, calcineurin inhibitors or incretin-based therapy which in the Investigator's opinion could interfere with glucose or lipid metabolism 90 days prior to screening
* Cancer (except basal cell skin cancer or squamous cell skin cancer) or any other clinically significant disorder, which in the investigator's opinion could interfere with the results of the trial
* Clinical suspicion of cardiac disease currently investigated
* Cardiac disease defined as: decompensated heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months
* Body mass index (BMI) <20 kg/m2 and/or >50 kg/m2
* Females of childbearing potential who are pregnant, breast-feeding, intend to become pregnant or are not using adequate contraceptive methods*
* Impaired liver function (transaminases > two times upper reference levels)
* The receipt of any investigational product 90 days prior to this trial
* Known or suspected abuse of alcohol or narcotics
* Screening calcitonin ≥ 50 ng/l
* Subjects with personal or family history of medullary thyroid carcinoma or a personal history of multiple endocrine neoplasia type 2

Lawfully detained, institutionalised and patients who are unable to give informed consent due to physical or mental conditions will not be included.

* Intrauterine devices and hormonal contraceptives (oral pills, patches, implants, vaginal rings, and injections) are considered as adequate contraceptives. Females of childbearing potential must use one of these contraceptives throughout the entire study plus 1 week after last injection with study medication. Surgical sterile (by bilateral vasectomy, tubectomy, hysterectomy or oophorectomy) or postmenopausal (defined as amenorrheic for at least one year) female participants are not considered as having a childbearing potential and are not required to use contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Plasma glucose during oral glucose tolerance test at week 26 | The trial visit of week 26
  Difference between the two treatment arms in plasma glucose concentrations during a 3h 75g-OGTT on the trial visit of week 26

SECONDARY OUTCOMES:
Hypoglycemic incidents | From the randomisation to trial visit of week 26
  Total hypoglycemic episodes during intervention
Fasting values of glucometabolic hormones | The trial visit of week 26
  Fasting plasma glucose, proinsulin, insulin and glucagon
Insulin resistance | The trial visit of week 26
  Insulin resistance evaluated by homeostasis model assessment (HOMA)
Beta cell function | The trial visit of week 26
  Beta-cell function evaluated by HOMA
Change in glycemic state | The trial visit of week 26
  Change in glycemic state following oral glucose tolerance test (normal glucose tolerance (NGT, fasting plasma glucose < 6.1 mmol/l and 2h plasma glucose < 7.8 mmol/l), impaired fasting glucose (IFG, fasting plasma glucose ≥ 6.1 and < 7.0 mmol/l), impaired glucose tolerance (IGT, 2h plasma glucose ≥ 7,8 and < 11.1 mmol/l) and diabetes mellitus (DM, fasting plasma glucose ≥ 7 mmol/l or 2h plasma glucose ≥ 11.1 mmol/l))
Blood pressure | The trial visit of week 26
  Blood Pressure
Pulse | The trial visit of week 26
  Resting pulse
Weight | The trial visit of week 26
  Weight
Body composition | The trial visit of week 26
  Body composition by dual energy x-ray absorptiometry (DXA) scan
Cardiac function and perfusion | The trial visit of week 26
  Cardiac function and perfusion evaluated by Rb-PET/CT scan
Cardiac autonomic function | The trial visit of week 26
  Cardiac autonomic function evaluated by heart rate variability
Arterial stiffness | The trial visit of week 26
  Arterial stiffness evaluated by Augmentation index from Pulse wave analysis
Cardiovascular and endothelial risk markers | The trial visit of week 26
  Cardiovascular and endothelial risk markers (troponin T, troponin I, creatine kinase-MB, high-sensitivity C-reactive protein (hsCRP), plasminogen activator inhibitor 1 (PAI-1), Tissue plasminogen activator (tPA), urat, von Willebrand factor (vWF), vascular endothelial cell adhesion molecule (VCAM), intercellular adhesion molecule (ICAM), TNFalpha, proBNP, E-selectin and asymmetric dimethylarginine)
Prothrombotic state | The trial visit of week 26
  Prothrombotic state (fibrinogen, activated partial thromboplastin time (APTT) and thromboelastography (TEG))
Lipid profile | The trial visit of week 26
  Lipid profile
Plasma liraglutide | The trial visit of week 26
  Plasma liraglutide

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feldt-Rasmussen, Prof,MD,DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Nephrology, Rigshospitalet, Copenhagen, Denmark